CLINICAL TRIAL: NCT01761500
Title: Improve the Survival Rate of Chinese Children and Adolescents With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-Fei Sun, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ped-No-1
Record Dates: First submitted 2012-12-21; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Childhood Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's lymphoma;; Childhood and adolescence;; Survival Rate
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Modified BFM-90 protocol (Other): Using the Modified BFM-90 protocol to treat Chinese children and adolescents with NHL
  Interventions: Other: Modified BFM-90 protocol

INTERVENTIONS:
Other: Modified BFM-90 protocol — Using Modified BFM-90 protocol to treat Chinese children and Adolescents with NHL

SUMMARY:
Non-Hodgkin's lymphoma is an aggressive malignance disease in children and adolescents. This study was designed to evaluate the efficacy and toxicity of the modified NHL-BFM-90 protocol in Chinese children and adolescents with Non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Non-Hodgkin's Lymphoma (NHL) in children and adolescents include Burkitt's lymphoma (BL), diffuse large B cell lymphoma (DLBL), anaplastic large cell lymphoma (ALCL) and lymphoblastic lymphoma (LBL). These subtypes of NHL are an aggressive group of diseases. At present, in developed countries, 80 to 90% of children with NHL are cured by intensive, risk-adapted chemotherapy.The best protocols include BFM-90, LMB-89 and FAB/LMB/96. However, in developing countries, such as those with low and moderate incomes, the limited availability of resources is an obstacle for using these complicated and intensive protocols.As such, very simple protocols, such as the CHOP protocol, were often used to treat children and adolescents with NHL, thus resulting in poor survival rates. To improve the survival rate of Chinese children and adolescents with NHL, This study was designed to evaluate the efficacy and toxicity of this modified NHL-BFM -90 protocol in Chinese children and adolescents with NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated children and adolescents with Non-Hodgkin's lymphoma
2. Age ≤ 20 years
3. The informed consent of their guardians was obtained.

Exclusion Criteria:

1. Recurrence Non-Hodgkin's lymphoma
2. Age >20 years
3. No abide by the protocol

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 1998-03; Primary Completion 2008-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The event free survival (EFS) | Up to 5 years
  The event free survival (EFS) was defined as the time from the start of treatment to one of the following events: death from any cause, disease progression during treatment, relapse, or to the date of the last follow up if patient did not experience any event.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Up to 5 years
  To assess the number of adverse events from the start of treatment to one of the following events: death from any cause, disease progression during treatment, relapse, severe infection, therapy related complication and second malignancy.

OTHER OUTCOMES:
the characteristics of Chinese children and adolescents with NHL | Up to 5 years
  To assess and compare the characteristics of Chinese children and adolescents with NHL with that in western countries,such as sex, age, pathological subtypes,tumor involvement location and treatment outcome,and so on.